CLINICAL TRIAL: NCT06055933
Title: Acute Effect of Kinesio Taping and Extracorporeal Shock Wave Therapy on Pain Severity and Lower Extremity Functionality in Plantar Fasciitis
Brief Title: Effect of Kinesio Taping and Extracorporeal Shock Wave Therapy on Plantar Fasciitis
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Abdulkadir dağbaşı, physiotherapist, Necmettin Erbakan University
Other Study IDs: ADagbasi001
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Plantar Fasciitis
Keywords: Plantar fasciitis; extracorporeal shock wave therapy; ESWT; placebo ESWT; plantar fascia; Kinesio Taping
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ESWT: To the ESWT group, with the ESWT device (BTL-6000SWT, UK); Extracorporeal shock wave therapy at 10Hz frequency, 2.5 Barr energy and 2000 shock/session values was applied with a 15 mm head in a single session. Shock waves were applied directly to the most sensitive point detected in the medial of the calcaneus.
- Placebo ESWT: The placebo ESWT group was given the ESWT device sound recorded from the external audio device and the application was performed without the ESWT device operating.
- ESWT+KT: With ESWT device (BTL-6000SWT, UK); Extracorporeal shock wave therapy at 10Hz frequency, 2.5 Barr energy and 2000 shocks/session was applied in a single session with a 15 mm head. Shock waves will be applied directly to the most sensitive point detected in the medial calcaneus, then a tape consisting of 96% cotton and 4% lycra, water-resistant, porous and adhesive, 5 cm wide and 0.5 mm thick will be used. Taping will be done after the ESWT session and the tape will be asked to remain for a week.

SUMMARY:
Type of this study: Prospective randomized controlled study. Purpose: The aim of this study is to compare the acute effect of pain level, lower extremity functionality level and plantar fascia flexibility in patients with plantar fasciitis receiving Exportacorporeal Shock Therapy (ESWT).

To compare the acute effect of pain level, lower extremity functionality level and plantar fascia flexibility in patients with plantar fasciitis who received KT application in addition to ESWT treatment.

To compare the acute effect of pain level, lower extremity functionality level and plantar fascia flexibility in patients with plantar fasciitis receiving placebo application.

90 volunteers will be included in the study as ESWT (n=30), placebo ESWT (n=30), ESWT and KT (n=30) application groups. How effective is ESWT, ESWT and Kinesiotape versus placebo ESWT acutely in the treatment of plantar fasciitis?

DETAILED DESCRIPTION:
Plantar fasciitis is a common disease in athletes and the sedentary population, accompanied by pain and limitation of foot function. Hot-cold tampon application, nonsteroidal anti-inflammatory drug, heel cushion, night splint, plantar fascia and Achilles stretching exercise, kinesio taping (CT), ultrasound, and extracorporeal shock wave therapy are the methods used in the treatment of plantar fasciitis. The aim of this study is to compare the acute effect on pain level, lower extremity functionality and plantar fascia flexibility in patients with plantar fasciitis receiving ESWT, patients with plantar fasciitis receiving Kinesiotape in addition to ESWT, and patients with plantar fasciitis receiving placebo ESWT.

Age (years), height (cm) and body weight (kg) measured with an adult scale with a mechanical height measure, gender, occupation, affected side and dominant side of patients diagnosed with plantar fasciitis will be recorded.

Patients will be divided into three groups: ESWT (Group 1), ESWT and KT (Group 2), and Placebo/Sham (Group 3) application groups. ESWT (BTL-6000SWT, UK); A single session will be applied at 10 Hz frequency, 2.5 Barr energy and 2000 shocks/session.

For KT application, a tape consisting of 96% cotton, 4% lycra, water-resistant, porous and adhesive, 5 cm wide and 0.5 mm thick will be used. Taping will be done after the ESWT session and the tape will be asked to remain for a week. After the first examination of the physical therapy and rehabilitation specialist physician in the placebo/Sham group, the patient will be listened to the sound of the device through the audio device and ESWT application will be applied without the device working.

For clinical follow-up of the patients, visual pain scale (VAS) score, lower extremity functional scale score will be used before and one week after treatment, and plantar fascia flexibility will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult cases aged 18-65 years diagnosed with plantar fasciitis by a physical medicine and rehabilitation specialist,
* Cases willing to continue the study,
* In the anamnesis, cases with severe pain when taking the first step after waking up in the morning or after a long period of inactivity and progressive aggravation of the pain as the activity continues,
* Cases whose consent forms were obtained by being informed about the study.

Exclusion Criteria:

* Cases who have undergone foot and ankle surgery,
* Loss or decrease of sensation in the foot and ankle region for various reasons,
* Difficulty in communication that prevents treatment and evaluations from being carried out effectively,
* Pregnancy,
* Presence of local infection,
* Having a widespread or regional tumoral disease,
* Having circulatory disorders in the lower extremities, bleeding,
* Anticoagulant use,
* Application of other treatment methods such as cold/hot application, exercise, orthosis use, electrotherapy agents,
* Cases with a history of systemic, inflammatory, neurological or vascular disease.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers with a diagnosis of plantar fasciitis and meeting inclusion criteria
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | baseline, post treatment (at 1th week)
  ). VAS, with numbers from 0 to 10 on a 10 cm horizontal line; 0 means "no pain"; It was stated to the patients that 10 represented "unbearable pain". The degree of pain was recorded numerically between 0 and 10

SECONDARY OUTCOMES:
Lower Extremity Functional Scale | baseline, post treatment (at 1th week)
  Lower Extremity Functional Scale; It is a scale developed to evaluate individuals' lower extremity functions, skills and activity limitations, translated into Turkish, and its validity and reliability have been established. Scoring is made between 0-80, with higher values indicating better functional level.

OTHER OUTCOMES:
Plantar Fascia Elasticity Measurement | baseline, post treatment (at 1th week)
  The person will be asked to pull his/her fingers back without bending his/her knees and keeping the heel and metatarsal heads in contact with the wall, and the distance between the thumb and the wall will be measured in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Doğan, Principal Investigator — Necmettin Erbakan University; abdulkadir dağbaşı, Study Chair — Necmettin Erbakan University; Aynur Başaran, Study Chair — Karamanoğlu Mehmetbey University
Locations (1):
- Necmettin Erbakan Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided